CLINICAL TRIAL: NCT04016363
Title: Impact of the ProbeFix on the Workflow of Pharmacological Stress Echocardiography Examinations: a Prospective, Randomized Controlled Open Label Study
Brief Title: Impact of the ProbeFix on the Workflow of Pharmacological Stress Echocardiography Examinations
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Industrial partner was not able to provide funding
Sponsor: Amir Abbas Mahabadi (Other)
Responsible Party: Sponsor-Investigator, Amir Abbas Mahabadi, Principal Investigator, University Hospital, Essen
Organization: University Hospital, Essen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-TEMP815870-BO
Record Dates: First submitted 2019-07-08; First posted 2019-07-11 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProbeFix arm (Experimental): The echocardiography probe is fixated on the patient's thorax using the ProbeFix
  Interventions: Other: ProbeFix
- Controll arm (Active Comparator): The sonographer manually holds the probe on the patient's thorax
  Interventions: Other: Manual hold

INTERVENTIONS:
Other: ProbeFix — ProbeFix vs. manual hold of the ultrasound probe during pharmacological stress-echocardiography examinations
  Arms: ProbeFix arm
Other: Manual hold — ProbeFix vs. manual hold of the ultrasound probe during pharmacological stress-echocardiography examinations
  Arms: Controll arm

SUMMARY:
Pharmacological stress-echocardiography examinations are routinely performed in daily clinical practice. Usually, the echo probe is manually placed on the patient's thorax by the physician. The ProbeFix is a novel device, enabling the fixation of the ultrasound probe on the patient's thorax. Therefore, there is no need to manually hold the probe. This may improve the standardization of the examination and my reduce its duration. The present trial will investigate, whether the utilization of the ProbeFix reduces the duration of stress-echocardiography examinations and improves standardization of image acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing clinically indicated pharmacological stress-echocardiography
* Willingness to participate

Exclusion Criteria:

* Pharmacological stress echocardiography indication other than evaluation of stress induced ischemia (e.g. Low-Flow-Low-Gradient aortic valve stenoseis)
* poor image quality
* Early termination of the stress-echocardiography examination for clinical reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration of stress-echocardiography examination | During the examination
  Duration from start of dobutamine infusion to end of stage IV of dobutamine infusion

SECONDARY OUTCOMES:
Echocardiography axis deviation in 4 chamber view | During the examination
  In 3-dimensional 4-chamber view, the deviation of the axis as compared to baseline will be assessed

OTHER OUTCOMES:
Cost-effectiveness | During the examination
  Assessment of cost-effectiveness, comparing a potential benefit in exam duration with costs of the ProbeFix

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided